CLINICAL TRIAL: NCT00914277
Title: Randomized, Double-blind, Placebo and Active Controlled Study of the Activity of SAR407899A Single-dose on the Ability to Increase Duration of Penile Rigidity, Under Experimental Condition, in Patients With Mild to Moderate Erectile Dysfunction (ED).
Brief Title: SAR407899 Single-dose in Treatment of Mild to Moderate Erectile Dysfunction
Acronym: RHOKET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: International Clinical Development Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT10775; EudraCT:2009-009936-56
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Erectile Dysfunction
Keywords: Rho-kinase inhibitor; male impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Experimental): Period 1: placebo
  Period 2: sildenafil
  Period 3: SAR407899 dose level 2
  Period 4: SAR407899 dose level 1
  Interventions: Drug: SAR407899; Drug: Placebo; Drug: Sildenafil
- Sequence 2 (Experimental): Period 1: sildenafil
  Period 2: SAR407899 dose level 1
  Period 3: placebo
  Period 4: SAR407899 dose level 2
  Interventions: Drug: SAR407899; Drug: Placebo; Drug: Sildenafil
- Sequence 3 (Experimental): Period 1: SAR407899 dose level 1
  Period 2: SAR407899 dose level 2
  Period 3: sildenafil
  Period 4: placebo
  Interventions: Drug: SAR407899; Drug: Placebo; Drug: Sildenafil
- Sequence 4 (Experimental): Period 1: SAR407899 dose level 2
  Period 2: placebo
  Period 3: SAR407899 dose level 1
  Period 4: sildenafil
  Interventions: Drug: SAR407899; Drug: Placebo; Drug: Sildenafil

INTERVENTIONS:
Drug: SAR407899 — Oral administration
Drug: Placebo — Oral administration
Drug: Sildenafil — Oral administration

SUMMARY:
The primary objective of this clinical trial is to study the ability of SAR407899 to increase the duration of penile erection in male patients with mild-moderate Erectile Dysfunction.

The secondary objectives of this clinical trial are to study the ability of SAR407899 to shorten increase the time to erection duration of penile erection in male patients with mild-moderate Erectile Dysfunction and to determine the overall safety and tolerability of SAR407899 in these patients.

ELIGIBILITY:
Inclusion Criteria:

* male with mild to moderate erectile dysfunction for at least 6 months
* written informed consent

Exclusion Criteria:

* diabetes mellitus
* orthostatic hypotension
* hypogonadal testosterone level

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Duration of penile rigidity during sexual stimulation | 4 hours following drug administration

SECONDARY OUTCOMES:
Time to onset of penile rigidity | 4 hours following drug administration
Blood pressure | 12 hours following drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Lionel HOVSEPIAN, MD, Principal Investigator — SGS Aster Life Science Services - Paris-France
Locations (1):
- Sanofi-Aventis Administrative Office, Paris, France